CLINICAL TRIAL: NCT06431477
Title: A Multi-center, Randomized, Open-label, Active Comparator-controlled, Phase 4 Clinical Trial To Evaluate the Efficacy and Safety of Telmisartan Compared With Losartan in Patients With Diabetic Nephropathy and Hypertension
Brief Title: Efficacy and Safety of Telmisartan Compared With Losartan
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B115_02HT/DN2201
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Nephropathies; Hypertension
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension | interventions — Telmisartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan tablet (Experimental)
  Interventions: Drug: telmisartan
- Losartan tablet (Active Comparator)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: telmisartan — QD, PO
  Arms: Telmisartan tablet
Drug: Losartan — QD, PO
  Arms: Losartan tablet

SUMMARY:
A study to evaluate the efficacy and safety of telmisartan compared with losartan in patients with diabetic nephropathy and hypertension

DETAILED DESCRIPTION:
A Multi-center, Randomized, Open-label, Active comparator-controlled, Phase 4 Clinical Trial To Evaluate the Efficacy and Safety of Telmisartan Compared with Losartan in Patients with Diabetic Nephropathy and Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Male of Female subjects aged ≥19 or <75
* Type II Diabetes Mellitus subjects who have been taken medicine
* Subjects who have voluntarily decided to participate in this clinical trial and Signed ICF

Exclusion Criteria:

* Subjects with Type I Diabetes Mellitus
* Subjects with Primary hyper-aldosteronism
* Subjects with a history of drug or alcohol abuse or suspected patient within 1 year as of the time of screening
* Pregnant women, lactating women, or subjects who do not agree to use appropriate contraception during the clinical trial period
* Subjects who received other clinical trial drugs within 28 days of screening visit
* Subjects who are unable to participate in this clinical trial at the discretion of the investigator.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change rate from baseline in Spot-UACR(Albumin/Creatinine Ratio) | 24 weeks after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: BeomSeok Kim, M.D, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No